CLINICAL TRIAL: NCT00244257
Title: Phase I, Open-Label, Multi-center, Single-Dose, Dose-Escalating, Safety, Tolerability, Immunogenicity, Pharmacokinetics and Pharmacodynamic Study of GMA161 in Patients With Idiopathic Thrombocytopenic Purpura (ITP)
Brief Title: Safety Study of GMA161 in Patients With Idiopathic Thrombocytopenic Purpura (ITP)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to low enrollment.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMA16100104; NCT00245999 (obsolete NCT alias)
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: idiopathic thrombocytopenia purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — GMA-161

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Cohort 1
  Interventions: Biological: GMA161
- 2 (Experimental): Cohort 2
  Interventions: Biological: GMA161
- 3 (Experimental): Cohort 3
  Interventions: Biological: GMA161
- 4 (Experimental): Cohort 4
  Interventions: Biological: GMA161
- 5 (Experimental): Cohort 5
  Interventions: Biological: GMA161

INTERVENTIONS:
Biological: GMA161 — 0.1 mg/kg, IV infusion on Day 0 and monitored for 7 days with collection of blood samples
  Arms: 1
Biological: GMA161 — 0.3 mg/kg, IV infusion on Day 0 and monitored for 7 days with collection of blood samples
  Arms: 2
Biological: GMA161 — 0.6 mg/kg, IV infusion on Day 0 and monitored for 7 days with collection of blood samples
  Arms: 3
Biological: GMA161 — 1.0 mg/kg, IV infusion on Day 0 and monitored for 7 days with collection of blood samples
  Arms: 4
Biological: GMA161 — 3.0 mg/kg, IV infusion on Day 0 and monitored for 7 days with collection of blood samples
  Arms: 5

SUMMARY:
This study is designed to investigate the safety of a single infusion of GMA161 in patients with idiopathic thrombocytopenic purpura, as well as, the way the drug enters and leaves the body. In addition, throughout the study, platelet counts and other blood cell numbers will be measured. NOTE: A decision was made to terminate this study in June 2008 due to low enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to any study-related procedures
* Chronic idiopathic thrombocytopenic purpura diagnosed for at least 6 months
* A platelet count of < 100,000/mm^3 on 2 determinations at least 6 weeks apart, including 1 determination within 7 days prior to initiating study treatment. Patients on a stable dose of corticosteroids for 2 weeks prior to study entry and with a platelet count of < 100,000/mm^3 may be enrolled
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1, with a life expectancy of at least 6 months

Exclusion Criteria:

* Women who are pregnant or lactating
* Women of childbearing potential unless using a medically acceptable contraceptive precaution with the use of spermicide or are sexually inactive
* Women who plan to become pregnant within 6 months after the screening phase
* Evidence of excessive bleeding requiring hospitalization within 6 weeks of study entry or a red cell transfusion within 6 weeks of study entry
* Absolute neutrophil count < 2,000/mm^3
* Total bilirubin > 2 mg/dL or alanine transaminase (ALT) or aspartate transaminase (AST) > 3 times the upper limit of normal ranges in the institutional laboratory
* Creatinine > 2 mg/dL
* History of drug-induced thrombocytopenia, marrow failure syndrome, such as aplastic anemia or myelodysplasia, or thrombocytopenia related to viral or bacterial infection
* Elevated (≥ 1.5 times the upper limit of normal range) prothrombin time (PT) or partial thromboplastin time (PTT) (other than related to a lupus anticoagulant or contact factor defect)
* Evidence of active bacterial infection or viral infection
* Active hemolysis that requires red cell transfusion within 6 weeks of study entry (Patients with evidence of concurrent autoimmune hemolysis [Evan's Syndrome] will be allowed)
* History of clinically significant cardiac or pulmonary disease
* History of cancer, other than: basal cell skin cancer, squamous cell skin cancer with no previous chemotherapy treatment or disease-free carcinoma in situ of the cervix, for a minimum of 5 years from the time of Screening
* HIV infection or acute or persistent hepatitis B and C viral infection (characterized by positive hepatitis B surface antigen (HBsAg), positive anti-hepatitis C virus [HCV] or polymerase chain reaction [PCR] assays for HCV)
* History of concurrent autoimmune disorders requiring systemic treatment for involvement of organ systems other than cytopenias or thyroid disease
* Treatment with cyclophosphamide, vincristine, rituximab, or any other monoclonal antibody within 12 weeks of study infusion
* Treatment with intravenous immunoglobulin (IVIg) within 2 weeks of study drug infusion or Rh(D) immune globulin intravenous within 4 weeks of study drug infusion
* Treatment with an agent, other than IVIg or corticosteroids, for ITP within 4 weeks of study entry. The dose level of corticosteroids may not be increased or decreased within 2 weeks of study entry
* Use of any investigational drug within 12 weeks before Screening
* Other pathology that might interfere with the assessment of the safety or efficacy of the test article or other clinically significant, uncontrolled medical condition that, in the Investigator's opinion, might interfere with the assessment or follow-up.
* Patients who have been splenectomized within 2 months of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Evaluate safety, tolerability and pharmacokinetics (PK) of single intravenous (IV) infusions of GMA161 in patients with idiopathic thrombocytopenic purpura (ITP) | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- United States (6):
  - Los Angeles, California
  - San Diego, California
  - Bethesda, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Cleveland, Ohio